CLINICAL TRIAL: NCT03470155
Title: Operative Mitralklappenrekonstruktion Bei Funktionellen Mitralklappenvitien Bei Reduzierter Systolischer Ventrikelfunktion
Brief Title: Operative Mitral Valve Reconstruction in Functional mv Insufficiency With Reduced Systolic Ventricle Function
Acronym: REFORM-MR
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: REFORM-MR
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Mitral Valve Insufficiency; Left Ventricular Systolic Dysfunction; Mitral Valve Prolapse
Keywords: annuloplasty mitral valve; reduced LV function
MeSH Terms: conditions — Mitral Valve Insufficiency; Ventricular Dysfunction, Left; Mitral Valve Prolapse | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- functional mitral insufficiency op: Patients with functional mitral insufficiency with restricted leaflet movement during systole (type IIIb Carpentier) undergoing operative reconstruction (mitral valve repair)
  Interventions: Procedure: mitral valve repair

INTERVENTIONS:
Procedure: mitral valve repair — operative reconstruction

SUMMARY:
Functional mitral insufficiency poses a challenge with regard to the optimal time of intervention, particularly because they are frequently associated with left ventricular (LV) dilation and reduced LV ejection fraction (EF). The registry will document the underlying pathology by using transthoracal echo cardiography (TTE) with analysis of common tenting parameters. OP strategies, data and outcomes will be documented, as well as follow-up data for echocardiography, quality of life and MACCE outcomes after 6 months, 1 and 2 years.

DETAILED DESCRIPTION:
Prospective enrolment of all patients with mitral valve insufficiency and restricted movement of leaflets during systole into a multicentric registry. Exact analysis of the underlying pathology using TTE with analysis of tenting parameters. In patients without contraindications, functional preoperative MRT to determine the functional reserve of ventricular function. Documentation of the quality of life of the patients using the SF12 questionnaire before and after intervention. Documentation of follow-up data (SF12, TTE, NT-pro BNP) at 6 months, 1 and 2 years. Development of operative strategies to improve long-term outcomes in patients with severe LV dilation (typically accompanied by function mitral insufficiency type IIIb).

ELIGIBILITY:
Inclusion Criteria:

* functional mitral valve insufficiency with reduced mobility of leaflets during systole (type IIIb) - effective regurgitation orifice area > 20 mm2 / regurgitant volume > 30 ml/beat
* left ventricular ejection fraction <= 50% and /or left ventricular end-diastolic diameter >= 60 mm
* tenting of the proximal and / or anterior mitral leaflets

Exclusion Criteria:

* prolaps of leaflets (type II mitral regurgitation)
* combination intervention with aortic valve repair or replacement
* re-operation at mitral valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting at participating hospitals with mitral valve dysfunction type III b who give written consent to participate in the registry
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
recurrent mitral valve insufficiency > grade 2 | 2 years
  see above

SECONDARY OUTCOMES:
MACCE | 1 year
  major adverse cardiovascular and cerebrovascular events
re-intervention at mitral valve | 2 years
  see above
device therapy (e. g. left ventricular auxiliary device or heart transplant) due to progressive heart failure | 2 years
  see above
cardiovascular mortality | 2 years
  see above
re-hospitalisation due to heart failure | 2 years
  see above

CONTACTS AND LOCATIONS:
Overall Officials: Evaldas Girdauskas, MD, Principal Investigator — Universitäres Herzzentrum Hamburg am UKE
Locations (6):
- Germany (6):
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Zentralklinik Bad Berka, Bad Berka
  - Charité - Klinik für kardiovaskuläre Chirurgie, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Klinik und Poliklinik für Herz- und Gefäßchirurgie am UHZ am UKE, Hamburg
  - Deutsches Herzzentrum München, München

IPD SHARING:
Plan to Share IPD: No
no IPD will be made available

REFERENCES:
- [Derived] Pausch J, Harmel E, Reichenspurner H, Kempfert J, Kuntze T, Owais T, Holubec T, Walther T, Krane M, Vitanova K, Borger MA, Eden M, Hachaturyan V, Bramlage P, Falk V, Girdauskas E. Subannular repair in secondary mitral regurgitation with restricted leaflet motion during systole. Heart. 2023 Aug 24;109(18):1394-1400. doi: 10.1136/heartjnl-2022-322239. PMID 37376817
- [Derived] Girdauskas E, Pausch J, Reichenspurner H, Kempfert J, Kuntze T, Owais T, Holubec T, Krane M, Vitanova K, Borger M, Eden M, Hachaturyan V, Bramlage P, Falk V. Subannular repair for functional mitral regurgitation with reduced systolic ventricle function: rationale and design of REFORM-MR registry. J Cardiothorac Surg. 2022 Dec 30;17(1):343. doi: 10.1186/s13019-022-02045-9. PMID 36581901